CLINICAL TRIAL: NCT01548703
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of BCI 838 in Healthy Adult Subjects
Brief Title: A Multiple Ascending Dose Study of BCI-838 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrainCells Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BCI-632-CL-003
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: metabotropic glutamate receptors 2 and 3; antagonist; mGluR; ketamine; BDNF; Depression; Major Depressive Disorder; Treatment Resistant Depression; Mood Disorder; Phase 1 safety, tolerability and pharmacokinetics study
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Mood Disorders | interventions — BCI-838

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCI-838 Dosing Arm 1 (Experimental): Ten subjects will be enrolled, 8 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838
- BCI-838 Dosing Arm 2 (Experimental): Ten subjects will be enrolled, 8 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838
- BCI-838 Dosing Arm 3 (Experimental): Ten subjects will be enrolled, 8 will receive BCI-838 and 2 will receive matching placebo.
  Interventions: Drug: BCI-838

INTERVENTIONS:
Drug: BCI-838 — BCI-838 100 mg or matching placebo administered once daily for 7 days
  Arms: BCI-838 Dosing Arm 1
Drug: BCI-838 — BCI-838 or matching placebo administered once daily for 7 days; the dose of BCI-838 will be determined based on the safety and PK data from the preceding dosing arm.
  Arms: BCI-838 Dosing Arm 2
Drug: BCI-838 — BCI-838 or matching placebo administered once daily for 7 days; the dose of BCI-838 will be determined based on the safety and PK data from the preceding dosing arm.
  Arms: BCI-838 Dosing Arm 3

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of BCI-838 and its metabolite BCI-632 in healthy male and female subjects.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability following oral administration of multiple doses of BCI-838 in healthy male and female subjects. The pharmacokinetic profile of multiple oral doses of BCI-838 in healthy male and female subjects will also be assessed. In addition, the pharmacodynamic effects of BCI-838 on the central nervous system using quantitative electroencephalogram analysis will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female healthy volunteers, 18-55 years of age
* Body Mass Index (BMI) between 18.0 to 30.0 kg/m2 inclusive
* Female subjects must have a negative pregnancy test at screening and admission. Females of childbearing potential (not at least 2 years postmenopausal or surgically sterile) must be using a reliable, medically acceptable form of contraception for at least 30 days prior to the screening visit and must agree to continue such use throughout the duration of the study and for 3 months after the final dose of study drug.
* Good general health as determined by medical history and physical examination with no clinically significant medical findings and no clinically relevant medical or surgical history and no acute or ongoing conditions within the past 30 days
* Able to participate and willing to give written informed consent and to comply with the study restrictions

Exclusion Criteria:

* Clinically significant medical abnormality, chronic disease or history or presence of significant pulmonary, gastrointestinal, metabolic, cardiac, hepatic, renal or neurological disorder
* History or current use of alcohol abuse or drug addiction
* Participation in a drug study within 60 days prior to drug administration.
* Participation in more than 3 other drug studies in the 10 months preceding the start of this study
* Donation or blood loss of more than 50 mL of blood within 60 days prior to the first drug administration. Donation of more than 1.5 liters of blood in the 10 months preceding the start of this study
* Illness within 5 days prior to drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  Safety will be evaluated by adverse events, vital signs, ECG, clinical labs, and physical exam.

SECONDARY OUTCOMES:
Cmax, tmax, t1/2 , AUC, CL/F, Vz/F, and Kel of BCI-838 and BCI-632 | predose, at specified timepoints during the 7-day dosing period, and at Day 10 (72 hours post-dose)
  The pharmacokinetics of BCI-838 and its metabolite BCI-632 will be completed by assessment of Cmax, tmax, t1/2 , AUC, CL/F, Vz/F, and Kel.
Quantitative EEG (qEEG) assessments | predose, and at specified timepoints during the 7-day dosing period
  The pharmacodynamic effects of BCI-838 on the central nervous system will be evaluated using quantitative electroencephalogram analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International, Zuidlaren, Netherlands